CLINICAL TRIAL: NCT04940949
Title: Interventional, Randomized, Double-Blind, Placebo-Controlled, Single-Ascending Dose Study Part Investigating the Safety, Tolerability, and Pharmacokinetic and -Dynamic Properties of Lu AF90103 and a Double-Blind, Cross-Over Study Part Investigating the Safety Profile After Infusion of Lu AF90103 at Two Rates to Healthy Men
Brief Title: A Study to Evaluate Lu AF90103 in Healthy Men
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated based on new safety data.
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 18907A
Record Dates: First submitted 2021-05-27; First posted 2021-06-28 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single Intravenous (IV) Dose of Lu AF90103 (Experimental): Participants will receive a single IV dose of Lu AF90103.
  Interventions: Drug: Lu AF90103
- Single IV Dose of Placebo (Placebo Comparator): Participants will receive a single IV dose of placebo matching to Lu AF90103.
  Interventions: Drug: Placebo
- 2 Single IV Doses of Lu AF90103 (Experimental): Participants will receive 2 single IV doses of Lu AF90103 separated by at least 5 days.
  Interventions: Drug: Lu AF90103

INTERVENTIONS:
Drug: Lu AF90103 — Lu AF90103 - powder for solution for infusion
  Arms: 2 Single IV Doses of Lu AF90103; Single Intravenous (IV) Dose of Lu AF90103
Drug: Placebo — Placebo - powder for solution for infusion
  Arms: Single IV Dose of Placebo

SUMMARY:
The purpose of this study is to investigate the safety and tolerability of Lu AF90103 and what the body does to Lu AF90103 after single doses of the drug administered directly into a vein.

DETAILED DESCRIPTION:
This study is the first-in-human (FIH) study with Lu AF90103. The study is divided in two parts, Part A and Part B.

Part A is an interventional, randomized, double-blind, sequential-group, placebo-controlled, single-ascending dose study to investigate the safety, tolerability, pharmacokinetics, and pharmacodynamics of Lu AF90103 in healthy men.

Part B is an interventional, randomized, double-blind, cross-over study to investigate the safety profile after administration of Lu AF90103 as an infusion at two different rates to healthy young men.

The dosage in Part B is guided by the cohorts in Part A and is a repetition of one of the doses from Part A.

The total study duration per participant from baseline to the end of follow-up will be maximum 11 days in Part A and 16 days in Part B.

ELIGIBILITY:
Inclusion Criteria:

* The participant is ≥18 and ≤45 years of age at the Screening Visit for Cohorts A1 to A6 (excluding cohort A2b) or ≥55 to ≤65 for participants in the CSF sampling Cohorts A2b and A7.
* The participant has body mass index (BMI) ≥18.5 kilograms (kg)/square meter (m^2) and ≤30 kg/m^2 and body weight ≥60 kilograms (kg) at the Screening Visit and at the Baseline Visit.
* The participant has a normal resting electroencephalogram (EEG) at Screening.
* The participant is, in the opinion of the investigator, generally healthy based on medical history, a physical examination, vital signs, an electrocardiogram (ECG), and the results of the clinical chemistry, haematology, urinalysis, serology, and other laboratory tests.

Exclusion Criteria:

* The participant has or has had any clinically significant immunological, cardiovascular, respiratory, metabolic, renal, hepatic, gastrointestinal, endocrinological, haematological, dermatological, venereal, neurological, or psychiatric disease or other major disorder.

Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-05-26 (Actual); Primary Completion 2021-11-23 (Actual); Study Completion 2021-11-23 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events | From dosing (Day 1) to Day 16
Maximum Observed Concentration (Cmax) of Lu AF90103 and AF88361 in Plasma and Cerebrospinal Fluid (CSF) | 0 (predose) up to 96 hours postdose on Day 1 to Day 5
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinity (AUC0-inf) of Lu AF90103 and AF88361 in Plasma and CSF | 0 (predose) up to 96 hours postdose on Day 1 to Day 5
Total Clearance (CL) of Lu AF90103 and AF88361 | 0 (predose) up to 96 hours postdose on Day 1 to Day 5
Amount of Lu AF90103 and Lu AF88361 Excreted in Urine | 0 (predose) up to 96 hours postdose on Day 1 to Day 5
Changes to Time Matched Baseline in Area Under the Curve (AUC) of Medial Prefrontal (FZ and CZ Electrodes) High Frequency Gamma Signal (100-170 Hertz [HZ]) for Lu AF90103 at the Resting State | From dosing (Day 1) to Day 4 (Part A) and Day 9 (Part B)
  The AUC of medial prefrontal (FZ and CZ electrodes) high frequency gamma signal (100-170 HZ) will be derived for Lu AF90103 at resting state, as measured by electroencephalogram (EEG).

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (1):
- QPS Netherlands B.V., GZ Groningen, Netherlands